CLINICAL TRIAL: NCT02132702
Title: Performance Attributes and User Progression While Using Ekso Robotic Exoskeleton in an Eight Week, Over Ground, Locomotor Program in Individuals With Spinal Cord Injury
Brief Title: Performance Attributes and User Progression While Using Ekso
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ekso Bionics (Industry)
Collaborators: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1-2013-082
Record Dates: First submitted 2014-05-02; First posted 2014-05-07 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

ARMS (1):
- Ekso treatment (Experimental)
  Interventions: Device: Ekso

INTERVENTIONS:
Device: Ekso

SUMMARY:
This study is to evaluate the performance attributes and user progression of participants with motor complete and incomplete spinal cord injury (SCI) while utilizing the Ekso robotic exoskeleton in an eight week over ground, locomotor program. We hypothesize an improvement in progression and overall health while using Ekso.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient or outpatient from 15 through 65 years of age at time of entry into the trial
* Motor complete (ASIA Impairment Scale [AIS] A and B), with a neurological level of injury (NLI) between C7-L2 (inclusive), or motor incomplete (AIS C and D), NLI C1-L2 (inclusive), as determined by the International Standards for Neurological Classification of SCI (ISNCSCI)
* Greater than 30 days since SCI occurred
* Height from 157 - 188 centimeters (5'2" to 6'2") or for individuals who do not meet this criteria the following criteria may be used as assessed per the Ekso operating manual:

Max hip width= 16.5" or 42cm Upper leg length= 20" to 24⅛" or 51cm to 61.4cm Lower leg length= 19" to 25" or 48cm to 63.4cm

* Maximum weight of 100 kilograms (220 pounds)
* Sufficient upper extremity (UE) strength to use a front wheeled walker (FWW) either by manual muscle testing (MMT) (minimum triceps strength bilaterally of 3/5, shoulder abduction/adduction and flexion/extension 4/5) and/or by functional standing test with FWW. Participants with impaired hand function may use cuff grips.
* Sufficient range of motion (ROM) to achieve a normal, reciprocal gait pattern, and normal sit to stand transitions.

  1. Hip extension greater than or equal to 5 degrees
  2. Knee extension greater than or equal to 5 degrees
  3. Ankle dorsiflexion greater than or equal to 0 degrees
* Demonstrate adequate trunk stability and upper extremity strength to utilize Ekso as evidenced by the ability to complete a level (or near level) surface wheelchair to mat transfer with minimal assistance.
* Medically stable and cleared by a physician for full weight bearing locomotor training including 15 minute standing frame trial to assess standing tolerance

Exclusion Criteria:

* Have trained in Ekso in the past except for one or two training/demonstration sessions
* Utilizing another robotic device for locomotor training
* Any medical issue that in the opinion of the Investigator precludes full weight bearing locomotor training including but not limited to:

  1. Spinal instability (or spinal orthotic unless cleared by physician)
  2. Acute deep vein thrombosis (DVT) with activity restrictions
  3. Severe, recurrent autonomic dysreflexia (AD) requiring medical intervention
  4. Heterotopic ossification (HO) in the lower extremities resulting in ROM restrictions at the hips or knees
  5. Two or more pathological fractures in the last 48 months in a major weight bearing bone (femur or tibia) in the lower extremity
  6. Hip subluxation (x-rays will be obtained for individuals injured prior to 10 years of age)
* Any medical issue that in the opinion of the Investigator would affect participant safety either due to cognitive deficits/impulsivity, intolerance to mild exercise or other factors
* Any issue that in the opinion of the Investigator would confound results such as a concurrent neurological injury or disorder (other than SCI) or other factors
* Modified Ashworth Scale (MAS) = 4 in the majority of lower extremity joints (e.g. greater than or equal to four joint movements in bilateral lower extremities when testing hip flexion/extension, knee flexion/extension, ankle dorsi/plantar flexion)
* Skin integrity issues in areas that contact the device (including abdominal ostomies) or that would prohibit sitting
* Pregnancy

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fin Biering-Sorensen, MD, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (9):
- Glostrup Hospital, Hornbæk, Denmark
- Universitats-und Rehabilitationskliniken, Ulm, Germany
- Heliomare Revalidatie, Wijk aan Zee, Netherlands
- Sunnaas Sykehus HF, Oslo, Norway
- Spain (2):
  - Institut Guttmann, Neurorehabilitation Hospital, Barcelona
  - Fundacion Lesionado Medular, Madrid
- Sweden (2):
  - Clinical Department of Rehabilitation Medicine and Department of Medicine and Health Services, Linköping
  - Sinalenheten, Akademiska Sjukhuset, Uppsala
- Swiss Paraplegic Center (SPZ), Nottwil, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- Ekso Treatment: Ekso gait training 3x/week for 8 weeks. Utilized the EksoGT device for approximately 60 minutes per session
Period: Overall Study
Arm/Group | Ekso Treatment
Started | 60
Completed | 52
Not Completed | 8
Not completed — Protocol Violation | 2
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: 8 participants who did not complete the study were not included in data synthesis or analysis - for this reason, only 52 participants were included below, which is different from the 60 who began the study.
Groups:
- Ekso Treatment: Ekso gait training 3x/week for 8 weeks
Arm/Group | Ekso Treatment
Number analyzed (Participants) | 52
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 35.8 [27.5 to 52.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 36
Region of Enrollment [Number; unit: participants]
  Netherlands | 2
  Sweden | 10
  Norway | 4
  Denmark | 12
  Switzerland | 6
  Germany | 8
  Spain | 10
Body Mass Index (BMI) [Mean (Inter-Quartile Range); unit: kilogram/meters^2] | 24.1 [22 to 26.2]
Time since injury [Count of Participants; unit: Participants]
  Recently injured < or = 1 year | 25
  Chronically injured > 1 year | 27
Neurological level of injury (NLI) and severity of injury at baseline [Count of Participants; unit: Participants] — In participants with spinal cord injury, NLI refers to the most caudal/inferior segment of the cord with intact sensation and antigravity muscle function strength, provided that there is normal (intact) sensory and motor function rostrally/above. The American Spinal Injury Association impairment scale (AIS) is used to measure this and determine the completeness of injury which tells about sensation or function below that level. AIS D is separated because these patients are motor incomplete and therefore have a more positive prognosis.
  Participants
    C1-C4 AIS A, B, C | 0
    C5-C8 AIS A, B, C | 4
    T1-S5 AIS A, B, C | 29
    All AIS D | 19
Spinal cord injury aetiology [Count of Participants; unit: Participants]
  Sport/Leisure | 16
  Assault | 2
  Transport | 17
  Fall | 7
  Other traumatic cause | 1
  Non-traumatic spinal cord dysfunction | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Adherent to Gait Training Progression Using Ekso
Description: Participants were scheduled to utilize exoskeleton 3x per week for 8 weeks. The number of participants who completed this dose was tracked.
Time Frame: 24 sessions
Measure: Count of Participants; unit: Participants
Arm/Group | Ekso Treatment
Number analyzed (Participants) | 60
Participants | 52

2. Secondary Outcome: Cardiovascular Effect
Description: The heart rate and blood pressure while sitting, at rest, and during activity will be taken to measure cardiovascular health changes. The perceived rate of exertion will also be used to determine cardiovascular effect.
Time Frame: baseline (1st session), session #1, session #12, session #24, followup at 12 weeks. Sessions occur 3x/week over an 8 week training period with a follow up visit at week 12.
Population: Data not collected
Arm/Group | Ekso Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Impact of Ekso Training on Spasticity
Description: The impact of Ekso training on muscle spasticity will be measured using the Modified Ashworth Scale (MAS)
Time Frame: baseline (1st session), session #12, session #24, followup at 12 weeks. Sessions occur 3x/week over an 8 week training period with a follow up visit at week 12.
Population: Data not collected
Arm/Group | Ekso Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Timed Up and Go (TUG)
Description: Impact of Ekso training on gait in participants who are ambulatory prior to Ekso training will be evaluated while not wearing the exoskeleton. Participants evaluated are those with ambulatory abilities outside of Ekso and therefore can complete test. This ambulatory ability could have been present at baseline testing, or participants may have acquired walking ability during the course of this study. Participant begins in a standard arm chair sitting back, stands, walks 3 meters, turns around, walks back, and sits into the chair. The time it takes to complete this sequence of movements is tracked.
Time Frame: as for outcome 3
Population: Subset analysis based on data collection
Measure: Mean (95% Confidence Interval); unit: seconds
Groups:
- Recently Injured: Participants with injuries < or = to 1 year
- Chronically Injured Participants: Participants with injuries > 1 year
Arm/Group | Recently Injured | Chronically Injured Participants
Number analyzed (Participants) | 15 | 12
seconds
  Baseline | 38.3 [30.5 to 46.1] | 35 [21 to 49]
  Session 12 | 36.6 [29 to 44.2] | 31.4 [17.4 to 45.4]
  Session 24 | 31.3 [23.8 to 38.8] | 27.2 [13.2 to 41.2]
  Follow up | 28.3 [20.8 to 35.8] | 28.7 [14.7 to 42.6]

5. Secondary Outcome: Muscle Strength
Description: The muscle strength of each of 5 key lower extremity muscles on each leg will be analyzed on a scale of 0-5. Lower extremity muscle scores are then added together to give a full lower extremity muscle score with a minimum score of 0 and a maximum score of 50. For each muscle: 0=None; No visible or palpable contraction. 1=Trace; Visible or palpable contraction with no motion. 2=Poor; Full range of motion (ROM) gravity eliminated. 3=Fair; Full ROM against gravity. 4=Good; Full ROM against gravity, moderate resistance. 5=Normal; Full ROM against gravity, maximal resistance. Higher LEMS scores (closer to 50) indicate higher strength towards typical, unimpaired muscle strength. Scores that are lower, close to or at 0, indicate little to no strength in the lower extremities.
Time Frame: baseline (1st session), after session #1, session #12, session #24, followup at 12 weeks. Sessions occur 3x/week over an 8 week training period with a follow up visit at week 12.
Population: Sub analysis completed based on data collected
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Recently Injured | Chronically Injured Participants
Number analyzed (Participants) | 15 | 12
units on a scale
  Baseline | 19.4 [11.6 to 27.3] | 14.5 [7.7 to 21.3]
  Session 12 | 24.1 [16.3 to 32] | 14.8 [8 to 21.6]
  Follow up | 24 [16.1 to 31.8] | 14.7 [7.8 to 21.5]

6. Secondary Outcome: Change in Bladder Function
Description: Evaluate the function of bowel and bladder as impacted by Ekso training using Modified International SCI Lower Urinary Tract Basic Data Set
Time Frame: as for outcome 5
Population: Data not collected
Groups:
- Ekso Treatment: Ekso
Arm/Group | Ekso Treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Functional Abilities
Description: Functional abilities will be measured based on Spinal Cord Independence Measure II (SCIM II). This assessment is scored from 0-100 with higher numbers equating to higher function/ more independence.
Time Frame: baseline, session #12, session #24, followup at 12 weeks. Sessions occur 3x/week over an 8 week training period with a follow up visit at week 12.
Population: 8 total drop outs
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Recently Injured | Chronically Injured Participants
Number analyzed (Participants) | 25 | 27
score on a scale
  Baseline | 62 [51 to 73] | 73 [64 to 77]
  Session 24 | 70 [65 to 77] | 74 [68 to 81]
  Follow up | 73 [67.5 to 78] | 74 [71 to 78]

8. Secondary Outcome: Change in Bowel Function
Description: The effect of Ekso training on bowel function will be evaluated using Modified International SCI Bowel Function Basic Data Set
Time Frame: baseline (1st session), session #24, followup at 12 weeks. Sessions occur 3x/week over an 8 week training period with a follow up visit at week 12.
Population: Data not collected
Arm/Group | Ekso Treatment
Number analyzed (Participants) | 0

9. Secondary Outcome: Quality of Life - Satisfaction of Life
Description: The Quality of Life change due to Ekso training will be evaluated using the International SCI Quality of Life Basic Data Sheet. Scores are from 1-10 with 1= completely dissatisfied and 10=completely satisfied.
Time Frame: baseline (1st session),session #24, followup at 12 weeks. Sessions occur 3x/week over an 8 week training period with a follow up visit at week 12.
Population: 8 total dropouts
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Recently Injured | Chronically Injured Participants
Number analyzed (Participants) | 25 | 27
score on a scale
  Baseline | 5 [3 to 7] | 6 [5 to 7]
  Session 24 | 6 [4.5 to 8] | 7 [6 to 9]
  Follow up | 6 [4 to 8] | 8 [7 to 8]

10. Secondary Outcome: Berg Balance Scale (BBS) - Balance
Description: Impact of Ekso training on gait in participants who are ambulatory prior to Ekso training. Gait progression will be evaluated in individuals with motor incomplete SCI who are ambulatory outside of Ekso. They will utilize Berg Balance Scale (BBS) to measure balance. The BBS includes 14 tasks each scored from 0-4, and the point value given for each of the 14 items is then summed together to yield a final score. Total BBS scores are out of 56 possible points where the higher the score, the better the balance is and therefore the lower the risk of falls. Scores can range from 0 to 56. A score or <45/56 is a commonly used standard that indicates individuals may be at greater risk of falling
Time Frame: as for outcome 3
Population: Subset of total participants based on data collection
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Recently Injured | Chronically Injured Participants
Number analyzed (Participants) | 15 | 12
score on a scale
  Baseline | 25.4 [18.2 to 32.5] | 25 [12.4 to 37.6]
  Session 12 | 28.8 [21.8 to 35.8] | 27.8 [15.2 to 40.4]
  Session 24 | 31.5 [24.6 to 38.4] | 28.9 [16.3 to 41.5]
  Follow up | 33.3 [26.4 to 40.2] | 29 [16.4 to 41.6]

11. Secondary Outcome: 10 Meter Walk Test - Gait Speed
Description: Impact of Ekso training on gait in participants who are ambulatory prior to Ekso training. Gait progression will be evaluated in individuals with motor incomplete SCI who are ambulatory outside of Ekso. They will utilize a 10 Meter Walk Test to analyze gait speed. Participants will walk over a 10 meter strip and the time taken to complete this is recorded.
Time Frame: as for outcome 3
Population: Subanalysis completed based on data collected
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Recently Injured | Chronically Injured Participants
Number analyzed (Participants) | 15 | 12
seconds
  Baseline | 35.3 [26.5 to 44.1] | 33.8 [20.8 to 46.8]
  Session 12 | 35.8 [27.1 to 44.4] | 33.2 [20.2 to 46.2]
  Session 24 | 28.6 [20 to 37.1] | 27.3 [14.3 to 40.3]
  Follow up | 26 [17.5 to 34.4] | 27 [14 to 40]

12. Secondary Outcome: Gait Progression
Description: Impact of Ekso training on gait in participants who are ambulatory prior to Ekso training. Gait progression will be evaluated in individuals with motor incomplete SCI who are ambulatory outside of Ekso. They will utilize the Walking Index for Spinal Cord Injury II (WISCI II) and note any changes in walking assistive device utilized. Scores on the WISCI II range from 0 to 20. A higher score indicates the participant can walk more independently (from braces, assistive device, and hands on assistance) whereas a lower score indicates that a participants requires assistance from a brace, assistive device, and/or another person.
Time Frame: as for outcome 3
Population: Subset analysis based on full data collection
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Recently Injured | Chronically Injured Participants
Number analyzed (Participants) | 15 | 12
units on a scale
  Baseline | 12.5 [10.5 to 14.4] | 14 [10.7 to 17.3]
  Session 12 | 12.6 [10.7 to 14.6] | 14.3 [11 to 17.6]
  Session 24 | 12.8 [11 to 14.7] | 13.7 [10.4 to 17]
  Follow up | 13.7 [11.8 to 15.5] | 13.9 [10.6 to 17.2]

ADVERSE EVENTS:
Time Frame: Study duration of 8 weeks plus 4 weeks of follow up
Groups:
- Ekso Treatment: Ekso gait training 3x/week for 8 weeks. While outcome measures were assessed in two groups, Recently Injured and Chronically Injured, adverse events were measured in one group out of all total participants because all participants underwent the same intervention (ie this one a 1-arm study)
Arm/Group | Ekso Treatment
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 22/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ekso Treatment (N=60)
Ankle swelling (Musculoskeletal and connective tissue disorders) | 3 (3)
dizziness or sycope (Cardiac disorders) | 8 (8)
Neurological symptoms (Nervous system disorders) | 3 (3)
Skin issues (Skin and subcutaneous tissue disorders) | 9 (9)
Concurrent medical issues (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No